CLINICAL TRIAL: NCT06372197
Title: Low-Income Group Psilocybin Assisted Therapy for Depression: A Feasibility Study
Brief Title: Low-Income Group Psilocybin Assisted Therapy for Depression
Acronym: LIGPATD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Hicks (Other)
Responsible Party: Sponsor-Investigator, Matthew Hicks, Principial Investigator, National University of Natural Medicine
Organization: National University of Natural Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIGPATD
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: poverty; low-income; psychedelics; psilocybin
MeSH Terms: conditions — Depression | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): This is an uncontrolled feasibility study with only one arm.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Following Oregon Psilocybin Services (OPS) rules, participants will be placed in cohorts of five to six, which whom they will do two 90-minute preparation session, two psilocybin sessions, and two 90-minute integration sessions. All sessions will be guided by two licensed facilitators.

SUMMARY:
Due to psilocybin-assisted therapy's success in previous research, growing cultural awareness and use of psilocybin and other psychedelics, the Oregon Psilocybin Services Act passed by ballot measure in 2020 and began offering services in 2023. While the program has had many successes, a significant problem it faces is affordability and no research to date has investigated the therapy in a low-income population.

Psychedelic research in recent decades has used the model of two therapists to one client to demonstrate an abundance of caution and safety to regulators, but no evidence has demonstrated this model to be safer or more effective than one with less practitioner oversight. This feasibility study would be the first investigation of Oregon Psilocybin Services as a model of care and among the first few to use a group therapy model. This study aims to test the feasibility of the model by assessing recruitment, retention, acceptability and safety of the treatment. In addition to an appropriate medical screening and intake the following questionnaire data will be collected: the Adverse Childhood Events (ACE) questionnaire, Credibility/Expectancy Questionnaire (CEQ), Hamilton Depression Inventory, PROMIS-29, Altered States of Consciousness (11-ASC) rating scale, and a survey and structured interview.

Participants will consist of adults in Oregon with an income at or below 200% of the federal poverty level. Inclusion criteria will include DSM-5 diagnosis of major depression. Participants will be individually screened by a study investigator and placed into groups of five to six participants. Treatment will consist of two group preparation sessions, two psilocybin sessions, and two group integration sessions. An additional follow-up visit to collect further data will take place three months after conclusion of the treatment.

The proposed study will provide valuable information for designing future clinical trials investigating the efficacy, mechanisms, and cost-effectiveness of psilocybin-assisted group therapy for depression in low-income populations.

ELIGIBILITY:
Inclusion Criteria:

* Oregon resident - this is due to the use of telehealth services and licenses of the study clinicians and their scope of practice within the state.
* Age 21 or older - Oregon Psilocybin Services Act sets the minimum eligible age of 21.
* Income 200% or below the Federal Poverty Line - this is the criteria for Oregon Medicaid (OHP).
* DSM-5 diagnosis of Major Depression Disorder.
* Current engagement with psychotherapy - no less than six therapy sessions in the previous six months and an intention to continue seeing their therapist no less than once every two weeks during the study period. This is to ensure participants have adequate psychological support during the study period. Participants must be willing to sign a release of information allowing study clinicians to communicate with their therapists.
* At least six months of stable housing history.
* Able to attend all study events.
* Able to read and speak fluent English.

Exclusion Criteria:

* A personal or family history of an immediate family member of schizophrenia, psychosis of any kind, mania, or hypomania.
* A current prescription for lithium.
* Active suicidal ideations or history of suicide attempts. Passive ideation, such as "I wouldn't mind if I never woke up again" is permissible.
* Uncontrolled hypertension.
* Any form of personality disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility | Beginning at study approval and funding through full enrollment, up to 18 months
  Determine the recruitment rate (number of participants enrolled compared to those approached) for low-income adults with depression into a group psilocybin-assisted therapy program.
Retention Feasibility | From participant enrollment through follow-up, up to 18 months
  Evaluate the participant retention rate throughout the study, including psilocybin sessions and follow-up assessments.
Acceptability | Assessed at the three month follow-up visit after completion of intervention
  Assess participant satisfaction with the group psilocybin-assisted therapy format through qualitative interviews and survey, including "On a scale of 0 to 5, zero being very dissatisfied and 5 being very satisfied, how would you rate your satisfaction with the treatment overall?"
Preliminary Safety and Tolerability: incidence and severity of adverse events | Through study completion, up to 18 months
  The incidence and severity of adverse events associated with psilocybin administration in a group setting will be documented and reported on to assess safety and tolerability.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Baseline (enrollment), integration #1 (3rd week of treatment), integration #2 (4th week of treatment), and follow-up (3 months post-treatment)
  Patient-Reported Outcomes Measurement Information System provides metrics for seven health related domains including depression.
Altered State of Consciousness rating scale (11-ASC) | At the end of both psilocybin sessions (week 3 and week 4).
  Provides a rating of intensity of altered state experiences across eleven domains.
Hamilton Depression Inventory | Baseline (enrollment), integration #1 (3rd week of treatment), integration #2 (4th week of treatment), and follow-up (3 months post-treatment)
  Provides a rating of depressive symptoms across several subdomains.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Hicks, ND, MS, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No